CLINICAL TRIAL: NCT02373566
Title: A Phase 2, Intra-patient Randomised Controlled Multicentre International Study to Evaluate the Efficacy of an Acellular Dermal Template Novomaix for the Treatment of Full Thickness Skin Defects
Brief Title: A Study to Evaluate the Efficacy of an Acellular Dermal Template for the Treatment of Full Thickness Skin Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Ernst Reichmann Tissue Biology Research Unit, Zürich (Other); Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESG-NVM-II-2014; NL50542.094.14 (Other: ABR)
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Full Thickness Skin Defects
Keywords: burns; dermal substitute; scar quality; reconstruction; wound healing; wound closure
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: part of wound treated with /without dermal template
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and assessor are both unaware of location of dermal template
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermal substitute with STSG (Experimental): Novomaix dermal substitute in combination with STSG
  Interventions: Device: Novomaix dermal substitute in combination with STSG
- STSG alone (No Intervention): STSG alone

INTERVENTIONS:
Device: Novomaix dermal substitute in combination with STSG — Novomaix dermal substitute in combination with STSG
  Other Names: Novomaix
  Arms: Dermal substitute with STSG

SUMMARY:
In this study the efficacy of an acellular dermal template (Novomaix), combined with split thickness skin grafts, for use in patients with full thickness skin defects, is tested. Results will be compared intra-patient with those obtained after conventional treatment with split thickness skin grafts. The investigators expect this treatment to provide better outcome regarding scar quality.

DETAILED DESCRIPTION:
Using dermal substitutes in combination with a split-thickness skin graft (STSG) is a well acknowledged therapy in burns and reconstructive surgery. Nevertheless, the ideal substitute is not available yet. We therefore want to investigate the use of an acellular dermal template (Novomaix), in combination with STSG, to treat these defects. Patients with with full thickness skin defects will be included in this study. This phase II study aims to investigate the efficacy of the use of this dermal matrix, with regard to scar quality as determined for elasticity at 3 months after treatment. Moreover, graft take (5-7 days after treatment), epithelialisation (5-7 days and 2-3 weeks), and scar quality (3 and 12 months after treatment, as determined for elasticity, colour/pigmentation, and using a subjective scar assessment scale) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (for Zurich: ≤ 18 years)
* Full thickness skin defects configured in such a way that two comparable and measurable areas can be grafted, both of minimally 3x3 cm
* ≤ 50% TBSA full thickness skin defects at time of intervention
* Informed consent by the patient and/or legal representatives.

Exclusion Criteria:

* Patients with infected wounds
* Full thickness skin wounds located in face and/or genitals will not be included
* Pregnant or breast feeding females
* Patients with known concomitant medical conditions that may interfere with normal wound healing (e.g. immune deficiency, HIV, uncontrolled diabetes, treatment with corticoid therapy, collagenoses, cancer)
* Known allergy against porcine collagen or elastin
* Patients that are expected (according to the responsible medical doctor) to be non-compliant to the study protocol. (This includes patients with severe cognitive dysfunction/impairment and severe psychiatric disorders)
* Previous enrolment of the patient into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Scar quality as assessed for scar elasticity (experimental vs control area) as measured by Cutometer or as assessed using subjective scar assessment scale (POSAS) | 3 months post-operative
  Scar elasticity as measured by Cutometer or as assessed using subjective scar assessment scale (POSAS)

SECONDARY OUTCOMES:
Graft take (Subjective assessment by experienced observer) | 5-7 days
Epithelialisation (Subjective assessment by experienced observer) | 5-7 days and 2-3 weeks post-operative
  Subjective assessment by experienced observer
Scar quality (Scar elasticity as measured by Cutometer or as assessed using POSAS questionnaire) | 12 months
  Scar elasticity as measured by Cutometer or as assessed using POSAS questionnaire
Scar quality (As determined with subjective scar assessment scale (POSAS) | 3 and 12 months
  As determined with subjective scar assessment scale (POSAS)
Scar quality (As measured for scar colour and pigmentation using DSM II ColorMeter) | 3 and 12 months
  As measured for scar colour and pigmentation using DSM II ColorMeter

CONTACTS AND LOCATIONS:
Overall Officials: Esther Middelkoop, Prof. dr., Principal Investigator — Red Cross Hospital
Locations (3):
- Zentrum für Schwerbrandverletzte mit Plastischer Chirurgie, Berlin, Germany
- Red Cross Hospital, Beverwijk, North Holland, Netherlands
- Children's Hospital Department of Surgery Kinderspital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Boekema BK, Vlig M, Olde Damink L, Middelkoop E, Eummelen L, Buhren AV, Ulrich MM. Effect of pore size and cross-linking of a novel collagen-elastin dermal substitute on wound healing. J Mater Sci Mater Med. 2014 Feb;25(2):423-33. doi: 10.1007/s10856-013-5075-2. Epub 2013 Nov 1. PMID 24178984
- See also: euroskingraft results — https://cordis.europa.eu/article/rcn/125139/it